CLINICAL TRIAL: NCT05514028
Title: Evaluation of Salivary RNAs in the Presence of an Adnexal Mass of Ovarian Origin - OVAmiARN Study
Brief Title: Evaluation of Salivary RNAs in the Presence of an Adnexal Mass of Ovarian Origin
Acronym: OVAmiARN
Status: Recruiting | Type: Observational
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry); iGenSeq (Unknown)
Responsible Party: Sponsor
Other Study IDs: FR-22-01
Record Dates: First submitted 2022-07-04; First posted 2022-08-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer; Ovarian Cyst Benign; Borderline Ovarian Cancer
Keywords: Cancer; RNA; machine learning algorithms; Ovarian
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cyst Benign: 100 patients
  Interventions: Other: Salivary samples
- Ovarian Cancer: 120 patients
  Interventions: Other: Salivary samples
- Borderline Ovarian Cancer: 30 patients
  Interventions: Other: Salivary samples

INTERVENTIONS:
Other: Salivary samples — For patients with a benign ovarian cyst, 1 saliva sample taken at 3 times (concomitant with a visit performed in routine care):
  * During the inclusion visit,
  * At the postoperative visit,
  * At the 6-month follow-up visit
  For patients with ovarian cancer, 1 saliva sample taken at different times (concomitant with a visit performed in routine care):
  * At the inclusion visit,
  * During the postoperative visit,
  * At the follow-up visits (6 months post-surgery and then every 6 months until 24 months)
  For patients with a borderline ovarian tumor, 1 saliva sample taken at different times (concomitant with a visit performed in routine care):
  * At the inclusion visit,
  * During the postoperative visit,
  * During pre- and post-chemotherapy visits (before and after each cycle)
  * During follow-up visits (every 4 months until 24 months)

SUMMARY:
OVAmiARN is a multicentre, prospective, longitudinal, non-interventional, observational study carried out in 8 obstetrics and gynecology departments in France; in order to describe the evolution of salivary miRNA expression between the pre-operative and post-therapy visits according to the type of mass. In time, the clinical application will be to significantly reduce the time to diagnosis and improve the care pathway for ovarian adnexal mass.

The study population consists of patients with an ovarian adnexal mass diagnosed by clinical examination and imaging (pelvic ultrasound and/or MRI) and requiring surgical management in routine care.

The patients concerned by the study will be managed without modification of the care pathway, nor modification of the therapeutic indications, nor modification of the diagnostic or follow-up examinations (imaging or biology) necessary according to the context, which are carried out according to the recommendations of the HAS, CNGOF.

In this study, the management and follow-up of patients :

* Are not imposed by the study: the doctor remains free to make medical prescriptions (treatments and examinations) and to determine the interval between consultation visits,
* Are not modified in comparison with the usual follow-up, except for the performance of the Collection of saliva

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* A patient with an ovarian adnexal mass diagnosed by clinical examination and imaging and likely to be ovarian cancer, a borderline tumour or a benign cyst,
* Patient with an indication for surgery
* Patient has dated and signed the consent form,
* Patient affiliated to the healthcare system,

Exclusion Criteria:

* Pregnant patient
* Patient infected with human immunodeficiency virus (HIV),
* Patient with significant difficulties in reading or writing the French language.
* Patient with another diagnosed cancer
* Patient with a history of cancer less than 5 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with an ovarian adnexal mass diagnosed by clinical examination and imaging (pelvic ultrasound and/or MRI and/or blood tumour markers) and requiring surgical management in routine care.
  The patients concerned by the study already benefit from a surgical management in different gynecology-obstetrics/gynecological oncology departments in France, Canada and Tunisia, as well as from a validation of the therapeutic indications in accordance with the national practices in force.
  The patients concerned by the study will be managed without modification of the care pathway, nor modification of the therapeutic indications, nor modification of the diagnostic or follow-up examinations (imaging and/or blood tumour markers) necessary according to the context which are carried out according to the national and/or international recommendations in force.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the Receiver Operating Curve (ROC) | Through the end of study inclusions, an average of 6 months
  Identifying a signature of ovarian cancer diagnosis by analysis of coding and non-coding RNAs in the saliva of subjects

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de Caen, Caen, Calvados
  - CHU Angers, Angers
  - CH Bastia, Bastia
  - CHU Lyon Sud / Hospices Civils de Lyon, Lyon
  - Centre Antoine Lacassagne, Nice
  - CH Niort, Niort
  - CHU Tenon, Paris
  - CHU Rennes, Rennes
  - Clinique La sagesse, Rennes
  - CHU Rouen, Hôpital de Bois-Guillaume, Rouen
  - Clinique Pasteur, Toulouse
  - CHRU Bretonneau-Tours, Tours